CLINICAL TRIAL: NCT06968494
Title: Safety and Tolerability of a Novel Implantable Device for the Treatment of Erectile Dysfunction Following Radical Prostatectomy
Brief Title: Safety and Tolerability of a Novel Implantable Device for the Treatment of Erectile Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Comphya Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-1.103
Record Dates: First submitted 2025-04-10; First posted 2025-05-13 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Erectile Dysfunction Following Radical Prostatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Implanted group (Experimental): Participants in the implanted group will be implanted with the study device during ongoing prostatectomy surgery.
  Interventions: Device: Activation of pro-erectile nerves within the pelvic plexus
- Control group (No Intervention): Participants in the control group will undergo standard prostatectomy and will not be implanted with the study device.

INTERVENTIONS:
Device: Activation of pro-erectile nerves within the pelvic plexus — The study device is an active implantable device. The device activates the pro-erectile nerves by delivering electrical pulses. The daily delivery of electrical pulses to the pro-erectile nerves may allow participants to recover natural erectile function.
  Arms: Implanted group

SUMMARY:
The goal of this clinical trial is to assess if a new device is safe to use as a potential treatment for erectile dysfunction following radical prostatectomy.

The main questions it aims to answer are:

* Is the device safe?
* Does the device works well? Are the participants satisfied with the device?

Participants will be implanted with the device during the ongoing prostatectomy surgery and will be asked to complete the following tasks during 6 months follow-up:

* Come to the hospital for follow-up visits,
* Complete questionnaires,
* Activate the device every day,
* Measure erection hardness.

Researchers will compare an implanted group (participants having the device) with a control group (participants not having the device) to see if the device works well.

ELIGIBILITY:
Inclusion Criteria:

* Men of ages between 30-75 years with indication for nerve-sparing prostatectomy surgery;
* Cancer stage T1c and T2a;
* Grade Groups 1 and 2 as well as low volume Grade Group 3 (Gleason score 4 + 3 = 7), as determined by biopsy (2 cores or less GG3) or single index MRI lesion of GG3 disease;
* IIEF-15 erectile function domain score equal to or greater than 26;
* Men interested in minimizing the effect of radical prostatectomy on erectile function;
* Ability to read and understand patient information materials and willingness to sign a written informed consent.

Exclusion Criteria:

* Men with neurological disease, including a history of spinal cord injury or trauma;
* IIEF-15 erectile function domain score less than 26;
* Failure to demonstrate adequate nocturne erectile function prioi prostatectomy (nocturnal RigiScan measure);
* Men with PSA > 20 ng/mL;
* History of ED, priapism and Peyronie disease;
* History of previous pelvic surgery, trauma or irradiation therapy;
* Currently have an active implantable device.
* Patient diagnosed with neurologic degenerative diseases that may negatively impact erectile functions;
* Identification of technical or clinical limitation to properly apply the use of nerve-sparing techniques during operation;
* Inability to understand and demonstrate device use instructions;
* Patients with insulin-dependent diabetes who suffer peripheral neuropathy or other diabetes associated complications;
* Patient unwillingness to engage in sexual activity;
* Patient is currently participating in another clinical investigation that would serve as a contraindication to implant a neurostimulator device to augment erectile function;
* Have participated in any drug or device trial in the last 4 weeks or plan to participate in any other drug or device study during the next 24 months;
* Possess any other characteristics that, per the investigator's judgment, may increase the risk or impair data collection for the procedure/study;
* Patient is a member of a vulnerable population (Vulnerable participants include those who lack consent capacity, including the mentally ill, prisoners, cognitively impaired participants, and employee volunteers).

Ages: 30 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender eligibility: male. Not based on self-representation of gender identity.
Enrollment: 20 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events | 6 months
  Adverse events will be systematically reported.
Occurrence of surgical complications | 6 months
  Surgical complications will be ranked according to the Clavien-Dindo classification
Occurrence of device deficiencies | 6 months
  Device deficiencies will be systematically reported and recorded.
Pain assessment | 6 months
  Participants will be asked to rate pain on a visual analog scale (from 0 to 10)

SECONDARY OUTCOMES:
Device Effectiveness | 6 months
  Device effectiveness will be assessed by asking participants to complete validated questionnaires.
Erectile function rehabilitation | 6 months
  Nocturnal penile erections will be assessed with the RigiScan device. Nocturnal erections reflect the extent of rehabilitation of natural erectile function.
Duration of Surgical Implantation Procedure | During surgical procedure
  Time (in minutes) from initial implant placement to final suture of the implant.
Ease of Implantation Steps | During surgical procedure
  Surgeon-reported rating of the ease of each implantation step using a standardized ordinal scale.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Pavlovich, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States